CLINICAL TRIAL: NCT05355805
Title: A Phase 2b Study to Evaluate the Efficacy and Safety of Izokibep in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Hidradenitis Suppurativa Phase 2b Study of Izokibep
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACELYRIN Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21102; 2021-005713-13 (EudraCT Number)
Record Dates: First submitted 2022-04-12; First posted 2022-05-02 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-03

CONDITIONS: Hidradenitis Suppurativa
Keywords: hidradenitis suppurativa; Izokibep
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A (Open-label) izokibep every week (Experimental): Participants will receive izokibep every week from Day 1 through Week 31
  Interventions: Drug: Izokibep
- Part B (Double-blind) izokibep every week (Experimental): Participants will receive izokibep every week for 31 weeks.
  Interventions: Drug: Izokibep
- Part B (Double-blind) izokibep every other week (Experimental): Participants will receive izokibep every other week for 30 weeks.
  Interventions: Drug: Izokibep
- Part B (Double-blind) placebo every week (Placebo Comparator): Participants will receive placebo every week up to Week 15, then izokibep from Week 16 to Week 31.
  Interventions: Drug: Placebo to izokibep
- Part B (Double-blind) placebo every other week (Placebo Comparator): Participants will receive placebo every other week up to Week 14, then izokibep from Week 16 to Week 30.
  Interventions: Drug: Placebo to izokibep

INTERVENTIONS:
Drug: Izokibep — Biologic: IL-17A inhibitor
  Form: Solution for injection
  Route of administration: Subcutaneous (SC)
  Arms: Part A (Open-label) izokibep every week; Part B (Double-blind) izokibep every other week; Part B (Double-blind) izokibep every week
Drug: Placebo to izokibep — Form: Solution for injection
  Route of administration: Subcutaneous (SC)
  Arms: Part B (Double-blind) placebo every other week; Part B (Double-blind) placebo every week

SUMMARY:
Izokibep is a potent and selective inhibitor of interleukin 17A (IL-17A) that is being developed for treatment of hidradenitis suppurativa (HS).

This study will evaluate the efficacy, safety, and immunogenicity of izokibep administered subcutaneously (SC) in adult subjects with moderate to severe HS.

ELIGIBILITY:
Inclusion Criteria:

General

* Subject has provided signed informed consent including consenting to comply with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* 18 years to 75 years of age

Type of Subject and Disease Characteristics

* Diagnosis of hidradenitis suppurativa (HS) for ≥ 1 year prior to first dose of study drug.
* Hidradenitis suppurativa lesions present in ≥ 2 distinct anatomic areas, one of which is Hurley Stage II or III.
* A total abscess and inflammatory nodule (AN) count of ≥ 5 at screening and Day 1 prior to enrollment/randomization.
* Subject must have had an inadequate response to oral antibiotics OR exhibited recurrence after discontinuation to, OR demonstrated intolerance to, OR have a contraindication to oral antibiotics for treatment of their HS.
* Must agree to use daily over-the-counter topical antiseptics.
* Subject must be willing to complete a daily skin pain diary for at least 3 days prior to Day 1 visit.

Exclusion Criteria:

Medical Conditions

* Draining fistula count of > 20.
* Outpatient surgery ≤ 8 weeks prior or inpatient surgery ≤ 12 weeks prior to enrollment/randomization.
* Other active skin disease or condition that could interfere with study assessments.
* Chronic pain not associated with HS.
* Uncontrolled, clinically significant system disease.
* History of demyelinating disease or neurological symptoms suggestive of demyelinating disease.
* Malignancy within 5 years.
* The subject is at risk of self-harm or harm to others.
* Active infection or history of certain infections.
* Tuberculosis or fungal infection seen on available chest x-ray taken ≤ 3 months of screening or at screening (Exception: documented evidence of completed treatment and clinically resolved).
* Known history of human immunodeficiency virus (HIV).

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Betah, MD, Study Director — ACELYRIN Inc.
Locations (40):
- United States (19):
  - Clinical Research Site, Birmingham, Alabama
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Fountain Valley, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Ocala, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Sandy Springs, Georgia
  - Clinical Research Site, Savannah, Georgia
  - Clinical Research Site, Rolling Meadows, Illinois
  - Clinical Research Site, Indianapolis, Indiana
  - Clinical Research Site, Plainfield, Indiana
  - Clinical Research Site, Murray, Kentucky
  - Clinical Research Site, Baton Rouge, Louisiana
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Mason, Ohio
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Pittsburgh, Pennsylvania
  - Clinical Research Site, Webster, Texas
- Canada (5):
  - Clinical Research Site, London, Ontario
  - Clinical Research Site, Markham, Ontario
  - Clinical Research Site, Waterloo, Ontario
  - Clinical Research Site, Québec, Quebec
  - Clinical Research Site, Saskatoon, Saskatchewan
- Germany (4):
  - Clinical Research Site, Bad Bentheim, Lower Saxony
  - Clinical Research Site, Bochum, Northwest
  - Clinical Research Site, Kiel, Schleswig-Holstein
  - Clinical Research Site, Schwerin
- Hungary (2):
  - Clinical Research Site, Budapest, BU
  - Clinical Research Site, Debrecen, HB
- Poland (6):
  - Clinical Research Site, Krakow, Lesser Poland Voivodeship
  - Clinical Research Site, Wroclaw, Lower Silesian Voivodeship
  - Clinical Research Site, Bialystok, Podlaskie Voivodeship
  - Clinical Research Site, Katowice, Silesian Voivodeship
  - Clinical Research Site, Lublin
  - Clinical Research Site, Szczecin
- Spain (4):
  - Clinical Research Site, Palma de Mallorca, PM
  - Clinical Research Site, Pontevedra, PO
  - Clinical Research Site, Manises, V
  - Clinical Research Site, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at different centers in the United States, Canada, Germany, Hungary, Poland, and Spain, and participated from May 2022 to February 2024.
Pre-assignment Details: Part A was a single-arm, open-label, proof-of-concept investigation to explore preliminary efficacy and safety of izokibep.
  Once Part A was fully enrolled, subsequent participants were enrolled into Part B.
  Part B was a randomized, double-blind, placebo-controlled, parallel-group, dose-finding investigation to evaluate the efficacy, safety, and immunogenicity of izokibep in participants with moderate to severe hidradenitis suppurativa.
Groups:
- Part A Izokibep 160 mg QW (Open-label): Participants with moderate to severe Hidradenitis Suppurativa (HS) received open label izokibep 160 mg by subcutaneous (SC) injection once every week (QW) in Part A for up to 31 weeks.
- Part B Placebo QW/Q2W Then Izokibep QW/Q2W: Participants with moderate to severe HS received placebo by SC injection either QW or every 2 weeks (Q2W) up to 16 weeks. After Week 16, participants who received placebo QW switched to izokibep QW up to Week 31. Participants who received placebo Q2W switched to izokibep Q2W for up to Week 30.
- Part B Izokibep 160 mg QW: Participants with moderate to severe HS received izokibep 160 mg QW by SC injection for 31 weeks.
- Part B Izokibep 160 mg Q2W: Participants with moderate to severe HS received izokibep 160 mg Q2W by SC injection for 30 weeks.
Period: Overall Study
Arm/Group | Part A Izokibep 160 mg QW (Open-label) | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W
Started | 30 | 59 | 57 | 59
Switched to Izokibep 160 mg QW | 0 | 24 | 0 | 0
Switched to Izokibep 160 mg Q2W | 0 | 26 | 0 | 0
Completed | 17 | 34 | 31 | 40
Not Completed | 13 | 25 | 26 | 19
Not completed — Lost to Follow-up | 6 | 11 | 10 | 6
Not completed — Decision by Sponsor | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 14 | 15 | 13

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS), Part A: all participants who received at lease one dose of study drug in Part A.
  FAS, Part B: all participants randomized in Part B.
Groups:
- Part A Izokibep 160 mg QW: Participants with moderate to severe HS received open label izokibep 160 mg by SC injection QW in Part A for up to 31 weeks.
- Part B Placebo QW/Q2W Then Izokibep QW/Q2W: Participants with moderate to severe HS received placebo by SC injection either QW or Q2W for up to 16 weeks. After Week 16, participants who received placebo QW switched to izokibep QW up to Week 31. Participants who received placebo Q2W switched to izokibep Q2W up to Week 30.
- Total: Total of all reporting groups
Arm/Group | Part A Izokibep 160 mg QW | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W | Total
Number analyzed (Participants) | 30 | 59 | 57 | 59 | 205
Age, Categorical [Count of Participants; unit: Participants] — Population: Participants in Part A and Part B of the study were analyzed separately
  Participants
    Part A: number analyzed (Participants) | 30 | 0 | 0 | 0 | 30
    Part A: <=18 years | 0 |  |  |  | 0
    Part A: Between 18 and 65 years | 30 |  |  |  | 30
    Part A: >=65 years | 0 |  |  |  | 0
    Part B: number analyzed (Participants) | 0 | 59 | 57 | 59 | 175
    Part B: <=18 years |  | 0 | 0 | 0 | 0
    Part B: Between 18 and 65 years |  | 58 | 56 | 58 | 172
    Part B: >=65 years |  | 1 | 1 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants in Part A and Part B of the study were analyzed separately
  years
    Part A: number analyzed (Participants) | 30 | 0 | 0 | 0 | 30
    Part A | 38.3 (9.68) |  |  |  | 38.3 (9.68)
    Part B: number analyzed (Participants) | 0 | 59 | 57 | 59 | 175
    Part B |  | 37.2 (11.45) | 35.3 (11.66) | 40.3 (10.04) | 37.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants in Part A and Part B of the study were analyzed separately
  Participants
    Part A: number analyzed (Participants) | 30 | 0 | 0 | 0 | 30
    Part A: Female | 21 |  |  |  | 21
    Part A: Male | 9 |  |  |  | 9
    Part B: number analyzed (Participants) | 0 | 59 | 57 | 59 | 175
    Part B: Female |  | 40 | 39 | 36 | 115
    Part B: Male |  | 19 | 18 | 23 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants in Part A and Part B of the study were analyzed separately
  Participants
    Part A: number analyzed (Participants) | 30 | 0 | 0 | 0 | 30
    Part A: Hispanic or Latino | 4 |  |  |  | 4
    Part A: Not Hispanic or Latino | 26 |  |  |  | 26
    Part A: Unknown or Not Reported | 0 |  |  |  | 0
    Part B: number analyzed (Participants) | 0 | 59 | 57 | 59 | 175
    Part B: Hispanic or Latino |  | 9 | 11 | 7 | 27
    Part B: Not Hispanic or Latino |  | 50 | 46 | 52 | 148
    Part B: Unknown or Not Reported |  | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants in Part A and Part B of the study were analyzed separately
  Participants
    Part A: number analyzed (Participants) | 30 | 0 | 0 | 0 | 30
    Part A: American Indian or Alaska Native | 0 |  |  |  | 0
    Part A: Asian | 0 |  |  |  | 0
    Part A: Native Hawaiian or Other Pacific Islander | 0 |  |  |  | 0
    Part A: Black or African American | 14 |  |  |  | 14
    Part A: White | 16 |  |  |  | 16
    Part A: More than one race | 0 |  |  |  | 0
    Part A: Unknown or Not Reported | 0 |  |  |  | 0
    Part B: number analyzed (Participants) | 0 | 59 | 57 | 59 | 175
    Part B: American Indian or Alaska Native |  | 0 | 1 | 0 | 1
    Part B: Asian |  | 1 | 3 | 0 | 4
    Part B: Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 | 0
    Part B: Black or African American |  | 9 | 7 | 6 | 22
    Part B: White |  | 47 | 45 | 51 | 143
    Part B: More than one race |  | 2 | 1 | 2 | 5
    Part B: Unknown or Not Reported |  | 0 | 0 | 0 | 0
Abscess Count [Mean (Standard Deviation); unit: Abcesses] — Population: Participants in Part A and Part B of the study were analyzed separately
  Abcesses
    Part A: number analyzed (Participants) | 30 | 0 | 0 | 0 | 30
    Part A | 1.7 (2.18) |  |  |  | 1.7 (2.18)
    Part B: number analyzed (Participants) | 0 | 59 | 57 | 59 | 175
    Part B |  | 1.8 (2.10) | 1.9 (3.57) | 1.9 (4.86) | 1.9 (3.67)
Inflammatory Nodule Count [Mean (Standard Deviation); unit: Nodules] — Population: Participants in Part A and Part B of the study were analyzed separately
  Nodules
    Part A: number analyzed (Participants) | 30 | 0 | 0 | 0 | 30
    Part A | 8.8 (7.20) |  |  |  | 8.8 (7.20)
    Part B: number analyzed (Participants) | 0 | 59 | 57 | 59 | 175
    Part B |  | 7.5 (5.10) | 10.0 (8.45) | 7.9 (4.21) | 8.5 (6.22)
Draining Fistula Count [Mean (Standard Deviation); unit: Fistulas] — Population: Participants in Part A and Part B of the study were analyzed separately
  Fistulas
    Part A: number analyzed (Participants) | 30 | 0 | 0 | 0 | 30
    Part A | 1.7 (2.35) |  |  |  | 1.7 (2.35)
    Part B: number analyzed (Participants) | 0 | 59 | 57 | 59 | 175
    Part B |  | 3.5 (5.18) | 3.0 (3.97) | 2.6 (3.38) | 3.1 (4.24)
Abcess and Inflammatory Nodule (AN) Count [Mean (Standard Deviation); unit: Total Abcess/Nodules] — Population: Participants in Part A and Part B of the study were analyzed separately
  Total Abcess/Nodules
    Part A: number analyzed (Participants) | 30 | 0 | 0 | 0 | 30
    Part A | 10.5 (7.64) |  |  |  | 10.5 (7.64)
    Part B: number analyzed (Participants) | 0 | 59 | 57 | 59 | 175
    Part B |  | 9.3 (5.24) | 11.9 (9.50) | 9.9 (6.85) | 10.4 (7.42)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants Who Achieved Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) at Week 12
Description: HiSCR75 was defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining fistula count.
Time Frame: Part A: Baseline to Week 12
Population: FAS, Part A: all participants who received at lease one dose of study drug in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Izokibep 160 mg QW
Number analyzed (Participants) | 30
Participants | 12

2. Primary Outcome: Part B: Number of Participants Who Achieved HiSCR75 at Week 16
Description: as for outcome 1
Time Frame: Part B: Baseline to Week 16
Population: FAS, Part B: all participants randomized in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W
Number analyzed (Participants) | 59 | 57 | 59
Participants | 16 | 21 | 19
Statistical Analysis 1: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg QW; The common risk difference between placebo QW/Q2W and the izokibep 160 mg QW arm among the four strata, prior biologic/Janus Kinase (JAK) inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error was estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Non-response imputation was used for participants with missing HiSCR75; Test type: Superiority; p = 0.3055, Cochran-Mantel-Haenszel — The estimated risk difference divided by the standard error was used as the test statistic and a p-value calculated assuming that the test statistic follows a standard normal distribution under the null hypothesis; Risk Difference (RD) = 8.27, Standard Error of Mean 8.075
Statistical Analysis 2: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg Q2W; The common risk difference between placebo QW/Q2W and the izokibep 160 mg Q2W arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error was estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Non-response imputation was used for participants with missing HiSCR75; Test type: Superiority; p = 0.6192, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 4.19, Standard Error of Mean 8.427

3. Secondary Outcome: Part A: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) referred to any untoward medical occurrence in a clinical study participant, regardless of a causal relationship with the study treatment. TEAEs included any event occurring after the participant received the study treatment. Clinically significant changes in vital signs, electrocardiograms, and laboratory tests recorded after treatment administration were documented as TEAEs. Serious TEAEs (SAEs) were untoward medical occurrences after the first dose, irrespective of a causal link to the study treatment, that led to death, were life-threatening, required hospitalization or its prolongation, caused significant disability, resulted in congenital anomalies, or were considered other medically important events.
Time Frame: Part A: Screening (Day -28) to Follow-up (Week 45), for a total of 49 weeks
Population: Safety analysis set (SAS): all participants who received at lease one dose of study drug in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Izokibep 160 mg QW
Number analyzed (Participants) | 30
Participants
  Any TEAE | 26
  Serious TEAE | 2

4. Secondary Outcome: Part A: Number of Participants Testing Positive for Anti-drug Antibodies (ADAs)
Description: Blood samples were collected at different time points throughout the study.
Time Frame: Baseline, Week 16, Week 32, Week 39
Population: ADA Analysis Set: all participants who received at lease one dose of study drug and had both baseline ADA and at least one post-dose ADA measurement in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Izokibep 160 mg QW
Number analyzed (Participants) | 25
Participants
  Baseline | 12
  Week 16: number analyzed (Participants) | 18
  Week 16 | 11
  Week 32: number analyzed (Participants) | 18
  Week 32 | 15
  Week 39: number analyzed (Participants) | 18
  Week 39 | 17

5. Secondary Outcome: Part B: Number of Participants Who Achieved HiSCR90 at Week 16
Description: HiSCR90 was defined as at least a 90% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining fistula count
Time Frame: Part B: Baseline to Week 16
Population: FAS, Part B: all participants randomized in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W
Number analyzed (Participants) | 59 | 57 | 59
Participants | 9 | 15 | 12
Statistical Analysis 1: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg QW; The common risk difference between placebo QW/Q2W and the izokibep 160 mg QW arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Non-response imputation was used for participants with missing HiSCR90; Test type: Superiority; p = 0.1606, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 10.14, Standard Error of Mean 7.229
Statistical Analysis 2: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg Q2W; The common risk difference between placebo QW/Q2W and the izokibep 160 mg Q2W arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Non-response imputation was used for participants with missing HiSCR90; Test type: Superiority; p = 0.5116, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 4.79, Standard Error of Mean 7.294

6. Secondary Outcome: Part B: Number of Participants Who Achieved HiSCR100 at Week 16
Description: HiSCR100 was defined as at least a 100% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining fistula count.
Time Frame: Part B: Baseline to Week 16
Population: FAS, Part B: all participants randomized in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B Placebo QW/Q2W Then Izokibep QW/Q2W: Participants with moderate to severe HS received placebo by SC injection either QW or Q2W up to 16 weeks. After Week 16, participants who received placebo QW switched to izokibep QW up to Week 31. Participants who received placebo Q2W switched to izokibep Q2W up to Week 30.
Arm/Group | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W
Number analyzed (Participants) | 59 | 57 | 59
Participants | 7 | 15 | 11
Statistical Analysis 1: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg QW; The common risk difference between placebo QW/Q2W and the izokibep 160 mg QW arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Non-response imputation was used for participants with missing HiSCR100; Test type: Superiority; p = 0.0514, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 13.67, Standard Error of Mean 7.019
Statistical Analysis 2: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg Q2W; The common risk difference between placebo QW/Q2W and the izokibep 160 mg Q2W arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Non-response imputation was used for participants with missing HiSCR100; Test type: Superiority; p = 0.3322, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 6.56, Standard Error of Mean 6.764

7. Secondary Outcome: Part B: Number of Participants Who Achieved HiSCR50 at Week 16
Description: HiSCR50 was defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining fistula count
Time Frame: Part B: Baseline to Week 16
Population: FAS, Part B: all participants randomized in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W
Number analyzed (Participants) | 59 | 57 | 59
Participants | 22 | 26 | 26
Statistical Analysis 1: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg QW; The common risk difference between placebo QW/Q2W and the izokibep 160 mg QW arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Non-response imputation was used for participants with missing HiSCR50; Test type: Superiority; p = 0.3258, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 8.63, Standard Error of Mean 8.780
Statistical Analysis 2: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg Q2W; The common risk difference between placebo QW/Q2W and the izokibep 160 mg Q2W arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Non-response imputation was used for participants with missing HiSCR50; Test type: Superiority; p = 0.4068, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 7.28, Standard Error of Mean 8.775

8. Secondary Outcome: Part B: Percentage of Participants Who Experienced ≥ 1 Disease Flare Through 16 Weeks of Treatment
Description: A flare was defined as ≥ 25% increase in AN count with a minimum increase of 2 AN relative to baseline.
  Missing data of abscess and inflammatory nodules counts at scheduled visits are imputed assuming monotone missingness pattern. Predictors in the regression model for missing values at Week 4 are Baseline Hurley stage, baseline abscess count, baseline inflammatory nodule count, baseline draining fistula count, sex, race, age, body mass index (BMI) and prior Biologic/JAK inhibitor use for HS. Predictors in the regression model for missing values after Week 4 are all of these variables, plus counts of abscess, inflammatory nodule, and draining fistula at prior scheduled assessment. Missing flare values in both the placebo and izokibep groups are imputed using observed data from the placebo group only.
Time Frame: Part B: Day 1 through to Week 16
Population: FAS, Part B: all participants randomized in Part B.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W
Number analyzed (Participants) | 59 | 57 | 59
Percentage of participants | 22.32 [11.7 to 32.9] | 18.29 [8.43 to 28.1] | 14.93 [5.72 to 24.1]
Statistical Analysis 1: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg QW; The common risk difference between placebo QW/Q2W and the izokibep 160 mg QW arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Missing data of abscess and inflammatory nodules counts at scheduled visits are imputed assuming monotone missingness pattern; Test type: Superiority — Predictors in the regression model for missing values at Week 16 are Baseline Hurley stage, baseline abscess count, baseline inflammatory nodule count, baseline draining fistula count, sex, race, age, BMI and Prior Biologic/JAK inhibitor use for HS plus counts of abscess, inflammatory nodule, and draining fistula at prior scheduled assessment. Missing flare values in both the placebo and izokibep groups are imputed using observed data from the placebo group only; p = 0.3329, Cochran-Mantel-Haenszel — The estimated risk difference divided by the standard error will be used as the test statistic and a p-value calculated assuming that the test statistic follows a standard normal distribution under the null hypothesis; Risk Difference (RD) = -7.40, Standard Error of Mean 7.661
Statistical Analysis 2: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg Q2W; The common risk difference between placebo QW/Q2W and the izokibep 160 mg Q2W arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting. Missing data of abscess and inflammatory nodules counts at scheduled visits are imputed assuming monotone missingness pattern; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.5882, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 4.06, Standard Error of Mean 7.574

9. Secondary Outcome: Part B: Number of Participants With Hurley Stage II at Baseline Who Achieved AN Count of 0, 1, or 2
Description: The percentage of participants with baseline Hurley Stage II who achieved AN count of 0, 1, or 2 at Week 16.
  Hurley stages:
  Stage 1 - solitary or multiple, isolated abscess formation without scarring or sinus tracts Stage 2 - recurrent abscesses, single or multiple widely separated lesions, with sinus tract formation Stage 3 - diffuse or broad involvement, with multiple interconnected sinus tracts and abscesses.
Time Frame: Part B: Week 16
Population: FAS, Part B: all participants randomized in Part B, inclusive only of participants with Hurley Stage II at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W
Number analyzed (Participants) | 34 | 35 | 36
Participants | 15 | 18 | 14
Statistical Analysis 1: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg QW; The common risk difference between placebo QW/Q2W and the izokibep 160 mg QW arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting; Test type: Superiority; p = 0.5422, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 7.31, Standard Error of Mean 11.995
Statistical Analysis 2: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg Q2W; The common risk difference between placebo QW/Q2W and the izokibep 160 mg Q2W arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting; Test type: Superiority; p = 0.6569, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = -5.23, Standard Error of Mean 11.770

10. Secondary Outcome: Part B: Number of Participants Who Achieved at Least a 3-Point Reduction From Baseline in Numeric Rating Scale (NRS) in Patient Global Assessment of Skin Pain at Its Worst at Week 16 Among Participants With Baseline NRS ≥ 4
Description: The Patient Global Assessment of Skin Pain is a NRS that consists of scores from 0 to 10 with 0 indicating "no skin pain" and 10 indicating "pain as bad as you can imagine".
Time Frame: Part B: Baseline to Week 16
Population: FAS, Part B: all participants randomized in Part B who had a baseline NRS ≥ 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W
Number analyzed (Participants) | 31 | 29 | 29
Participants | 4 | 5 | 9
Statistical Analysis 1: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg QW; The common risk difference between placebo QW/Q2W and the izokibep 160 mg QW arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting; Test type: Superiority; p = 0.4031, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 7.48, Standard Error of Mean 8.951
Statistical Analysis 2: Comparison: Part B Placebo QW/Q2W Then Izokibep QW/Q2W vs Part B Izokibep 160 mg Q2W; The common risk difference between placebo QW/Q2W and the izokibep 160 mg Q2W arm among the four strata, prior biologic/JAK inhibitor use for HS (Yes/No) and Hurley Stage (II or III), used for randomization and associated standard error will be estimated by combining the observed risk differences using Cochran-Mantel-Haenszel weighting; Test type: Superiority; p = 0.0327, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 21.27, Standard Error of Mean 9.959

11. Secondary Outcome: Part B: Number of Participants With TEAEs of Special Interest
Description: Adverse events of special interest were adverse events in the following categories: candida infection, inflammatory bowel disease, suicidal ideation, malignancies, major cardiovascular and cerebrovascular events, tuberculosis, infections, cytopenias and hypersensitivity reactions.
Time Frame: Part B: Screening (Day -28) to Follow-up (Week 45), for a total of 49 weeks
Population: SAS: all randomized participants who received at least one dose of study drug in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B Placebo QW/Q2W (Up to Week 16): Participants with moderate to severe HS received placebo by SC injection either QW or Q2W for up to 16 weeks.
- Part B Izokibep 160 mg Q2W (Up to Week 16): Participants received izokibep Q2W in a blinded manor for 16 weeks.
- Part B Izokibep 160 mg QW (Up to Week 16): Participants with moderate to severe HS received izokibep 160 mg QW by SC injection for 16 weeks.
- Part B Placebo/Izokibep 160 mg QW (Week 16 to 31): Participants received izokibep QW in a blinded manor for weeks 16-31.
- Part B Placebo/Izokibep 160 mg Q2W (Week 16 to 30): Participants received izokibep Q2W in a blinded manor for weeks 16-30.
- Part B: Izokibep 160 mg QW (Week 16 to 31): Participants with moderate to severe HS received izokibep 160 mg QW by SC injection during weeks 16-31.
- Part B: Izokibep 160 mg Q2W (Week 16 to 30): Participants with moderate to severe HS received izokibep 160 mg Q2W by SC injection during weeks 16-30.
Arm/Group | Part B Placebo QW/Q2W (Up to Week 16) | Part B Izokibep 160 mg Q2W (Up to Week 16) | Part B Izokibep 160 mg QW (Up to Week 16) | Part B Placebo/Izokibep 160 mg QW (Week 16 to 31) | Part B Placebo/Izokibep 160 mg Q2W (Week 16 to 30) | Part B: Izokibep 160 mg QW (Week 16 to 31) | Part B: Izokibep 160 mg Q2W (Week 16 to 30)
Number analyzed (Participants) | 59 | 59 | 57 | 24 | 26 | 43 | 53
Participants | 4 | 2 | 1 | 1 | 2 | 0 | 2

12. Secondary Outcome: Part B: Number of Participants With TEAEs
Description: An AE referred to any untoward medical occurrence in a clinical study participant, regardless of a causal relationship with the study treatment. TEAEs included any event occurring after the participant received the study treatment. Clinically significant changes in vital signs, electrocardiograms, and laboratory tests recorded after treatment administration were documented as TEAEs. SAEs were untoward medical occurrences after the first dose, irrespective of a causal link to the study treatment, that led to death, were life-threatening, required hospitalization or its prolongation, caused significant disability, resulted in congenital anomalies, or were considered other medically important events.
Time Frame: Part B: Screening (Day -28) to Follow-up (Week 45), for a total of 49 weeks
Population: SAS: all randomized participants who received at least one dose of study drug in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Placebo QW/Q2W (Up to Week 16) | Part B Izokibep 160 mg QW (Up to Week 16) | Part B Izokibep 160 mg Q2W (Up to Week 16) | Part B Placebo/Izokibep 160 mg QW (Week 16 to 31) | Part B Placebo/Izokibep 160 mg Q2W (Week 16 to 30) | Part B: Izokibep 160 mg QW (Week 16 to 31) | Part B: Izokibep 160 mg Q2W (Week 16 to 30)
Number analyzed (Participants) | 59 | 57 | 59 | 24 | 26 | 43 | 53
Participants
  Any TEAE | 40 | 49 | 48 | 17 | 16 | 27 | 25
  Serious TEAE | 2 | 2 | 1 | 2 | 1 | 1 | 0

13. Secondary Outcome: Part B: Number of Participants Testing Positive for ADAs
Description: Blood samples were collected at different time points throughout the study.
Time Frame: Up to 39 weeks
Population: ADA Analysis Set: all participants who received at lease one dose of study drug and had both baseline ADA and at least one post-dose ADA measurement in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Placebo QW/Q2W Then Izokibep QW/Q2W | Part B Izokibep 160 mg QW | Part B Izokibep 160 mg Q2W
Number analyzed (Participants) | 54 | 54 | 53
Participants
  Baseline | 27 | 29 | 36
  Week 16: number analyzed (Participants) | 47 | 41 | 49
  Week 16 | 21 | 29 | 39
  Week 32: number analyzed (Participants) | 20 | 46 | 19
  Week 32 | 13 | 35 | 12
  Week 39: number analyzed (Participants) | 18 | 40 | 18
  Week 39 | 17 | 32 | 15

ADVERSE EVENTS:
Time Frame: Part A: Screening (Day -28) to Follow-up (Week 45), for a total of 49 weeks. Part B: Screening (Day -28) to Follow-up (Week 45), for a total of 49 weeks.
Description: SAS: all randomized participants who received at least one dose of study drug.
Groups:
- Part B Izokibep 160 mg QW - (Up to Week 16): Participants with moderate to severe HS received izokibep 160 mg QW by SC injection for 16 weeks.
Arm/Group | Part A Izokibep 160 mg QW | Part B Placebo QW/Q2W (Up to Week 16) | Part B Izokibep 160 mg QW - (Up to Week 16) | Part B Izokibep 160 mg Q2W (Up to Week 16) | Part B Placebo/Izokibep 160 mg Q2W (Week 16 to 30) | Part B Placebo/Izokibep 160 mg QW (Week 16 to 31) | Part B: Izokibep 160 mg Q2W (Week 16 to 30) | Part B: Izokibep 160 mg QW (Week 16 to 31)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/59 | 0/57 | 0/59 | 0/26 | 0/24 | 0/53 | 0/43
Serious Adverse Events (participants affected / at risk) | 2/30 | 2/59 | 2/57 | 1/59 | 1/26 | 2/24 | 0/53 | 1/43
Other Adverse Events (participants affected / at risk) | 25/30 | 25/59 | 43/57 | 34/59 | 10/26 | 14/24 | 9/53 | 13/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Izokibep 160 mg QW (N=30) | Part B Placebo QW/Q2W (Up to Week 16) (N=59) | Part B Izokibep 160 mg QW - (Up to Week 16) (N=57) | Part B Izokibep 160 mg Q2W (Up to Week 16) (N=59) | Part B Placebo/Izokibep 160 mg Q2W (Week 16 to 30) (N=26) | Part B Placebo/Izokibep 160 mg QW (Week 16 to 31) (N=24) | Part B: Izokibep 160 mg Q2W (Week 16 to 30) (N=53) | Part B: Izokibep 160 mg QW (Week 16 to 31) (N=43)
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1)
Colonic abscess (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Still's disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Izokibep 160 mg QW (N=30) | Part B Placebo QW/Q2W (Up to Week 16) (N=59) | Part B Izokibep 160 mg QW - (Up to Week 16) (N=57) | Part B Izokibep 160 mg Q2W (Up to Week 16) (N=59) | Part B Placebo/Izokibep 160 mg Q2W (Week 16 to 30) (N=26) | Part B Placebo/Izokibep 160 mg QW (Week 16 to 31) (N=24) | Part B: Izokibep 160 mg Q2W (Week 16 to 30) (N=53) | Part B: Izokibep 160 mg QW (Week 16 to 31) (N=43)
Injection site erythema (General disorders) | 12 (38) | 0 | 31 (59) | 23 (44) | 7 (12) | 12 (75) | 5 (15) | 3 (17)
Injection site pruritus (General disorders) | 8 (23) | 0 | 16 (30) | 7 (10) | 5 (5) | 5 (24) | 2 (3) | 2 (4)
Injection site swelling (General disorders) | 6 (19) | 0 | 9 (12) | 5 (6) | 2 (3) | 3 (20) | 3 (4) | 0
Injection site warmth (General disorders) | 5 (6) | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 4 (13) | 0 | 1 (7) | 1 (7) | 0 | 0 | 1 (1) | 0
Injection site pain (General disorders) | 3 (9) | 1 (14) | 3 (19) | 3 (3) | 2 (3) | 3 (21) | 1 (1) | 1 (7)
Injection site induration (General disorders) | 0 | 0 | 0 | 1 (1) | 2 (3) | 0 | 0 | 1 (2)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 | 1 (1) | 0
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 | 0 | 2 (2) | 0 | 1 (1) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 | 3 (3) | 1 (1) | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 8 (15) | 8 (13) | 6 (6) | 0 | 1 (1) | 0 | 5 (7)
Hypertension (Vascular disorders) | 2 (2) | 3 (4) | 0 | 1 (1) | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 3 (3) | 0 | 0 | 1 (1) | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 5 (6) | 9 (10) | 5 (5) | 1 (1) | 0 | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 0 | 6 (7) | 5 (6) | 2 (2) | 0 | 1 (1) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 (4) | 1 (1) | 1 (1) | 1 (2) | 0 | 1 (1) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 (2) | 3 (3) | 0 | 0 | 0 | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 0 | 0 | 1 (2) | 0 | 1 (1) | 2 (3) | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per Clinical Trial Agreements, sites may not publish study results without sponsor's written consent:

* sponsor has right to first publication
* after first publication, site may publish if sponsor is given 60 days to review for confidential/proprietary information
* if publication may impact sponsor rights (eg, a patent), sponsor may request 90-day delay
* if sponsor does not publish within 12 months after study end or confirms they will not, site may publish, subject to sponsor's rights above

DOCUMENTS (2):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT05355805/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT05355805/SAP_002.pdf